CLINICAL TRIAL: NCT05607264
Title: Kinesio Taping Technique Versus Virtual Reality in Rehabilitation of Patients With Chronic Shoulder Impingement Syndrome
Brief Title: Kinesio Taping Technique Versus Virtual Reality in Patients With Chronic Shoulder Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hend Ali Mohamed, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Hend_PhD_2022
Record Dates: First submitted 2022-11-01; First posted 2022-11-07 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Impingement Syndrome, Shoulder
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Kinsiotaping (Experimental): patients who received kinesiotaping plus conventional treatment for chronic shoulder impingement syndrome.
  Interventions: Other: Kinsiotaping; Other: Conventional treatment
- Virtual Reality training (Experimental): patients who received VR training plus conventional treatment for chronic shoulder impingement syndrome.
  Interventions: Other: Motion-controlled VR games; Other: Conventional treatment
- conventional treatment (Active Comparator): patients who received conventional treatment for chronic shoulder impingement syndrome only.
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Other: Kinsiotaping — Patients received the kinesiotaping over supraspinatus muscle and deltoid muscle, tape will be removed every three days and subjects will return back to the clinic to reapplication of tape again. Patients received the same therapeutic treatment 3 times/ week for four weeks. KT is air permeable and water resistant, allowing it to stay in place for three to five days.
  Arms: Kinsiotaping
Other: Motion-controlled VR games — Virtual Rehab utilizes the unique characteristics of Microsoft Kinects motion technology to track and capture the movements of the patients so that patients become immersed in a 3D environment where they interact with the game. Subjects will include in a supervised virtual reality exergaming program for shoulder movements for 4 weeks, 3 days per week and 10 minutes for session.
  Arms: Virtual Reality training
Other: Conventional treatment — patients received conventional treatment for chronic shoulder impingement syndrome only.

SUMMARY:
Purpose of the Study: to compare between the effect of kinesio taping technique versus virtual reality technique in rehabilitation of patients with chronic shoulder impingement syndrome.

DETAILED DESCRIPTION:
Rotator cuff disorders are considered to be among the most common causes of shoulder pain and disability encountered in both primary and secondary care, with subacromial impingement syndrome in particular being the most common disorder, resulting in functional loss and disability, of the shoulder.

There is a lack of literature about virtual reality exergaming in subjects with orthopedic problems.

To reduce UL impairment, new therapeutic approaches, such as constraint-induced movement therapy, robotic arm training, and virtual reality therapy (VRT), have been successfully employed over the last decade.

Kinesio taping is the increasingly popular method for preventing and treating sports injuries. The tape helps to maintain the joint position, increases the proprioceptive awareness, and assists in removal of exudates thereby reducing pain and improves the muscle function.

So as there is lag in literature regarding the best type of treatment for patients with chronic impingement syndrome so this study will be conducted to compare between kinesiotaping and virtual reality and to determine the best treatment for patients with chronic Shoulder Impingement Syndrome (SIS).

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients will be diagnosed with chronic shoulder impingement syndrome (who had supraspinatus tendinitis stage (II) 2. Ages 25-40 years 3. Both sexes will be included. 4. Patients complaint from limitation in the ROM in abduction flexion and external rotation.

  5. Patient complaint from pain and tendinitis in subacromial area more than 3 in VAS.

  6. All patients complaint from difficulties in joining ADL activities. 7. All patients will assign written consent form.

Exclusion Criteria:

Subjects with the following criteria will be excluded from the study:

1. Shoulder fracture or instability.
2. Previous shoulder surgery.
3. Arthritis of the glenohumeral or acromioclavicular joints.
4. Cervical radiculopathy
5. Patients with visual disorders.
6. Diabetic patients.
7. Balance and coordination disorders.
8. Tumor and breast cancer.
9. Major trauma.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Assessing the change in musculoskeletal disorders of the upper limbs | at baseline and after 4 weeks of intervention
  Assessment by using Disabilities of the Arm, Shoulder, and Hand Questionnaire (DASH). The DASH is a 30-item self-report questionnaire designed to assess musculoskeletal disorders of the upper limbs. Scoring the DASH 30-item disability/symptom section:
  1) Item responses range from 1 (e.g. no difficulty, not at all, not limited, none, strongly disagree) to 5 (e.g. unable, extremely, unable, strongly agree). Scoring the optional 2 4-item high performance sections: 1) Add values of each response, then divide by 4, subtract 1 and multiply by 25: [((sum of values/4) - 1)*25]. 2) Optional modules should not be scored if items are missing. Arabic version of DASH questionnaire will be used, Which is reliable and valid to be used for evaluating upper extremity work related injuries.
Assessing the change in pain intensity | at baseline and after 4 weeks of intervention
  Assessment by using visual analouge scale (VAS). It was used to assess the intensity of pain. Operationally a VAS is usually a horizontal line, l00 mm in length, anchored by word descriptors at each end. The patient marks on the line the point that they feel represents their perception of their current state. The VAS score is determined by measuring in millimeters from the left hand end of the line to the point that the patient marks.
Assessing the change in shoulder range of motion | at baseline and after 4 weeks of intervention
  Assessment by using Electro goniometer. It was used to measure shoulder ROM (flexion, abduction, internal rotation).
Assessing the change in muscle activity of Supraspinatus muscle | at baseline and after 4 weeks of intervention
  Assessment by using Electromyogram (EMG). It was used to measure muscle activity of Supraspinatus, infraspinatus, anterior and middle deltoid.

CONTACTS AND LOCATIONS:
Overall Officials: Hend Ahmed, Physiotherapist, Principal Investigator — Cairo University
Locations (1):
- Outpatient clinic, Faculty of Physical Therapy, Cairo University, Egypt., Dokki, Egypt

IPD SHARING:
Plan to Share IPD: Undecided